CLINICAL TRIAL: NCT00509171
Title: A Prospective Randomized Trial Investigating the Effect of a Novel Reamer-Irrigator-Aspirator on the Incidence of Fat Embolism and Respiratory Function During Intramedullary Nailing of Femoral Shaft Fractures
Brief Title: Effect of a Novel Reamer-Irrigator-Aspirator on the Incidence of Fat Embolism
Acronym: RIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Orthopaedic Trauma Association (Other); Synthes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-6-30-MAR-07; NCT00753376 (obsolete NCT alias)
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Embolism; Femoral Fractures
Keywords: embolism; femur fracture; lavage; TEE; reamer; IM nail
MeSH Terms: conditions — Embolism; Femoral Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Standard reamer (Active Comparator): Standard reamer
  Interventions: Device: Reamer Irrigator Aspirator
- 2-Use of the Reamer-Irrigator Aspirator (Active Comparator): Use of the Reamer-Irrigator Aspirator
  Interventions: Device: Reamer Irrigator Aspirator

INTERVENTIONS:
Device: Reamer Irrigator Aspirator — Use of standard reamer vs reamer irrigator-aspirator during IM nailing of tibial shaft fractures

SUMMARY:
The purpose of this study is to determine the effect on the incidence of fat emboli when using a Reamer-Irrigator Aspirator during reamed IM nail fixation of femoral shaft fractures

DETAILED DESCRIPTION:
The current practice of reaming the medullary canal for the fixation of femur fractures is recommended, however, there is an associated increase in the level of embolic events which confers morbidity and, occasionally, mortality.

The RIA is a single device which is able to ream the medullary canal, irrigate the canal and subsequently aspirate the reamed medullary contents in order to get rid of medullary fat and other contents responsible for these adverse embolic events.

A novel Reamer-Irrigator-Aspirator (RIA) (Synthes, Inc) will be evaluated in a randomized study, to determine its effect on the incidence of fat emboli events during reamed IM nail fixation of consecutive femoral shaft fractures as measured by intra-operative transesophageal echocardiogram and pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 16 to 65 years of age
* Skeletally mature
* Isolated, closed femoral shaft fracture (participant may also have sustained a distal radius/wrist, distal tibia/ankle, hand, and/or foot fractures for eligible inclusion)
* Fracture amenable to an antegrade I.M. nail
* Fracture amenable to insertion of a 12 mm RIA
* Fracture ≤ 48 hrs post injury
* Participant has a 'Thorax' Abbreviated Injury Score (AIS) of < 2
* Participant has a 'Head & Neck' AIS score of < 2
* Provision of informed consent

Exclusion Criteria:

* Fracture proximal to the lesser trochanter
* Open fracture
* Participant has a humeral, tibial, contralateral femoral, spinal,and/or pelvic fracture
* Pathological fracture
* Fractures > 48 hrs post injury
* Limited life expectancy due to significant medical co-morbidities
* Previous history of esophageal/gastric surgery
* Previous history of esophageal/gastric tumor
* Previous history of esophageal varices
* Medical contraindication to surgery

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy A Hall, MD, FRCSC, Principal Investigator — Unity Health Toronto; Emil Schemitsch, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1-Standard Reamer | 2-Use of the Reamer-Irrigator Aspirator
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Standard Reamer | 2-Use of the Reamer-Irrigator Aspirator | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Full Range); unit: years] | 39.2 [17 to 69] | 39.2 [17 to 67] | 39.2 [17 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Embolic Debris
Description: The differences in total emboli score (Embolism Grading Scal3) between the 2 experimental groups were analyzed with a 2-sample 2-tailed t test.
  Embolism Grading Scale:
  Amount: Amount of right atrium fill by echogenic particles none = 0 less than ½ = 1 more than ½ = 2 complete fill = 3 Duration: Duration of echogenesis during 1-minute video segment (seconds) none = 0 less than 5 seconds = 1 5-30 seconds = 2 over 30 seconds = 3
  Size: Diameter of largest echogenic particle (mm):
  none = 0 less than 5mm = 1 5-10mm = 2 larger than 10mm = 3 Percent: 0 =no fill
  1. = less than 66 %
  2. = greater than 66%
Time Frame: Duration of surgical procedure.
Population: Antegrade IM nailing of a femoral shaft fracture with standard reamers or the RIA device. All patients were monitored intraoperatively with a continuous TEE to assess embolic events in the right atrium. Total emboli score was measured when using the RIA device during the REAM
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1-Standard Reamer | 2-Use of the Reamer-Irrigator Aspirator
Number analyzed (Participants) | 11 | 11
score on a scale | 5.3 (1.81) | 4.05 (2.19)

ADVERSE EVENTS:
Arm/Group | 1-Standard Reamer | 2-Use of the Reamer-Irrigator Aspirator
Serious Adverse Events (participants affected / at risk) | 2/11 | 2/11
Other Adverse Events (participants affected / at risk) | 3/11 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Standard Reamer (N=11) | 2-Use of the Reamer-Irrigator Aspirator (N=11)
prolonged intubation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — prolonged intubation due to oxygen desaturation.
femoral neck fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-Standard Reamer (N=11) | 2-Use of the Reamer-Irrigator Aspirator (N=11)
hardware irritation (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) — local irritation near proximal locking screws, which resolved with locking screw removal
decrease in hemoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — decrease in hemoglobin requiring transfusion on day 2 postoperatively

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days